CLINICAL TRIAL: NCT04973280
Title: A Study to Evaluate the Effectiveness of the Additional Risk Minimisation Measures (aRMMs) for REBLOZYL Among Healthcare Professionals (HCPs) in the European Economic Area (EEA)
Brief Title: Study to Evaluate Additional Risk Minimisation Measures (aRMMs) for REBLOZYL Among Healthcare Professionals (HCPs)
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: ACE-536-MDS-005
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Myelodysplastic Syndromes; Beta-thalassemia
Keywords: REBLOZYL; Myelodysplastic Syndromes; Healthcare Professionals; Post-authorization safety study; Additional educational measures; Beta-thalassemia; Luspatercept
MeSH Terms: conditions — Myelodysplastic Syndromes; beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare Professionals (HCPs): The PASS will be conducted among HCPs in a representative sample of EEA countries where REBLOZYL is commercially available. A sample of HCPs from EEA countries who manage care for patients with certain haematologic conditions and who may/do prescribe REBLOZYL will be recruited from the target population of HCPs who were sent the REBLOZYL aRMMs in these countries. The final list of countries to be included may include 1) only countries where reimbursement has been sought and gained, 2) a geographically representative sample (e.g., northern, southern, eastern, and western EU Members States to the degree possible based on the first criteria), 3) a mixture of countries with higher and lower REBLOZYL usage, and 4) other feasibility considerations such as the ability to conduct direct-to-HCP non-market research studies.

SUMMARY:
This is a non-interventional post-authorization safety study (PASS) employing a cross sectional design to evaluate the effectiveness of the additional risk minimization measures (aRMMs) for REBLOZYL. A survey will be used to measure the knowledge and comprehension of the REBLOZYL aRMMs among European Economic Area (EEA) based healthcare professionals (HCPs). The PASS will be conducted among HCPs in a representative sample of EEA countries where REBLOZYL is commercially available, potentially including Austria, Germany, Italy, Norway, Sweden, the Netherlands, Poland, and Spain. Additional EEA countries may be included, as needed, based on commercial availability and reimbursement status.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals (HCPs) experienced in treatment of haematological diseases who may intend to prescribe REBLOZYL in the participating European countries and were on the target group for dissemination of the additional risk minimization measures (aRMMs).
* The HCP provides permission to share their responses in aggregate with European Medicines Agency (EMA) or National Competent Authorities (NCAs), if requested.

Exclusion Criteria:

* HCPs who previously participated in the cognitive pre-testing of the survey questionnaires to be used for the study.
* HCPs who have been direct employees of the marketing authorization holder (MAH), the EMA, or the study vendor within the past 5 years.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare Professionals (HCPs) who were part of the REBLOZYL aRMMs dissemination list and who practice in any of the participating EEA countries.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Knowledge that although there are no data from the use of REBLOZYL in pregnant women, studies in animals exposed to REBLOZYL have shown reproductive toxicity and embryo-fetal toxicity | Up to 3 months
  Calculated as the percentage of healthcare professionals (HCPs) who answer "True" to question 1A
Knowledge that women of childbearing potential (WCBP) who become pregnant during treatment with REBLOZYL should not continue REBLOZYL treatment even if they receive appropriate monitoring | Up to 3 months
  Calculated as the percentage of HCPs who answer "False" to question 1B
Knowledge that HCPs must counsel WCBP of the potential teratogenic risk of REBLOZYL | Up to 3 months
  Calculated as the percentage of HCPs who answer "True" to question 1C
Knowledge that for WCBP who become pregnant during treatment with REBLOZYL, the pregnancy outcome should be evaluated | Up to 3 months
  Calculated as the percentage of HCPs who answer "False" to question 1D
Knowledge that the use of REBLOZYL is contraindicated during pregnancy and in WCBP who are not using at least 1 highly effective method of contraception | Up to 3 months
  Calculated as the percentage of HCPs who answer "True" to question 1E
Knowledge of what information about contraception methods should be provided when counselling WCBP | Up to 3 months
  Calculated as the percentage of HCPs who answer "WCBP should use at least 1 highly effective method of contraception during treatment with REBLOZYL and for at least 3 months after stopping treatment" to question 2
Knowledge of how many pregnancy tests should be performed for WCBP before they start treatment with REBLOZYL | Up to 3 months
  Calculated as the percentage of HCPs who answer "A single pregnancy test must be performed and medically verified before starting treatment with REBLOZYL" to question 3
Knowledge of the frequency pregnancy tests should be repeated for WCBP who are receiving treatment with REBLOZYL | Up to 3 months
  Calculated as the percentage of HCPs who answer "At suitable intervals and medically verified as negative" to question 4
Knowledge that WCBP should be informed to report a pregnancy that occurs during treatment with REBLOZYL and should receive counselling if they become pregnant | Up to 3 months
  Calculated as the percentage of HCPs who answer "True" to question 5
Knowledge of how long after stopping treatment with REBLOZYL should WCBP be informed to report a pregnancy that occurs and should they receive counselling if they become pregnant | Up to 3 months
  Calculated as the percentage of HCPs who answer "Pregnancies that occur within 3 months after stopping REBLOZYL should be reported and participants should receive counselling" to question 6
Always providing WCBP with the REBLOZYL Patient Card | Up to 3 months
  Calculated as the percentage of HCPs who answer "Yes, always" to providing the REBLOZYL Patient Card to WCBP (question 10-A). The denominator for this variable is the n who answer question 10 (not the n who answer 10-A)
Composite knowledge for all 5 items in the core question set | Up to 3 months
  A composite endpoint calculated as the percentage of HCPs who answer: None of questions 1E, 2, 3, 4, and 10-A correctly; 1 of questions 1E, 2, 3, 4, and 10-A correctly; 2 of questions 1E, 2, 3, 4, and 10-A correctly; 3 of questions 1E, 2, 3, 4, and 10-A correctly; 4 of questions 1E, 2, 3, 4, and 10-A correctly; All 5 of questions 1E, 2, 3, 4, and 10-A correctly

SECONDARY OUTCOMES:
Awareness of the HCP Checklist | Up to 3 months
  Calculated as the percentage of HCPs who answer "Yes" to question 7
Read/reviewed the HCP Checklist | Up to 3 months
  Calculated as the percentage of HCPs who answer "Yes, all of it" or "Yes, some of it" to question 8
Use of the HCP Checklist prior to initiating treatment | Up to 3 months
  Calculated as percentages of HCPs who answer "Always" or "Sometimes" to question 9A
Use of the HCP Checklist at each subsequent administration | Up to 3 months
  Calculated as percentages of HCPs who answer "Always" or "Sometimes" to question 9B
Use of the HCP Checklist for at least 3 months after stopping treatment | Up to 3 months
  Calculated as percentages of HCPs who answer "Always" or "Sometimes" to question 9C
Primary source from which HCPs learned about the appropriate indication, contraindications and precautions for use, and potential risks for REBLOZYL | Up to 3 months
  Calculated as the percentage of HCPs who tick each source in question 11 (for example, percentage of HCPs that ticked the REBLOZYL summary of product characteristics (SmPC), etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Local Institutions, Vienna, Austria
- Local Institutions, Brussels, Belgium
- Local Institutions, Berlin, Germany
- Local Institutions, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html